CLINICAL TRIAL: NCT02101580
Title: Phase 1B Trial of ADI-PEG 20 Plus Nab-Paclitaxel and Gemcitabine in Subjects With Advanced Pancreatic Cancer
Brief Title: Ph 1B Trial With ADI-PEG 20 Plus Nab-Paclitaxel and Gemcitabine in Subjects With Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2013-002
Record Dates: First submitted 2014-03-25; First posted 2014-04-02 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Advanced Pancreatic Cancer
Keywords: argininosuccinate synthetase; arginine; arginine deiminase
MeSH Terms: interventions — ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADI-PEG 20 (Experimental)
  Interventions: Drug: ADI-PEG 20

INTERVENTIONS:
Drug: ADI-PEG 20

SUMMARY:
Assessment of safety and tolerability of ADI-PEG 20 plus nab-Paclitaxel and Gemcitabine in subjects with Advanced Pancreatic Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of pancreatic carcinoma (dose escalation and MTD expansion components).
2. Subjects in the dose-escalation component can have had up to 1 prior line of systemic therapy. Subjects with pancreatic carcinoma to be enrolled in the MTD expansion cohort must have untreated, measurable metastatic disease. Subjects for the MTD cohort may have received prior adjuvant gemcitabine or fluoropyrimidine based therapy in the adjuvant setting provided more than 6 months has elapsed following completion of adjuvant therapy.
3. Unresectable disease or subject refused surgery.
4. Progressive disease if treated with chemotherapy, radiotherapy, surgery or immuno-therapy. If prior radiation was given, the measurable disease should be outside the radiation port.
5. Measurable disease as assessed by RECIST 1.1 criteria (Appendix A).
6. Age ≥ 18 years.
7. ECOG performance status of 0 - 1.
8. No prior systemic therapy, immunotherapy, investigational agent, or radiation therapy within the last 4 weeks. Radiation therapy for symptomatic relief is allowed within the last 2 weeks.

Exclusion Criteria:

1. Serious infection requiring treatment with systemically administered antibiotics at the time of study entrance, or an infection requiring systemic antibiotic therapy within 7 days prior to the first dose of study treatment.
2. Serious underlying lung function abnormality due to the risk of fatal pneumonitis that was caused by the combination of Abraxane and gemcitabine
3. Grade 2 or higher neuropathy (CTCAE V4.0)
4. Prior treatment with nab-paclitaxel.
5. Pregnancy or lactation.
6. Expected non-compliance.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, or psychiatric illness, social situations that would limit compliance with study requirements.
8. Subjects who have had any anticancer treatment prior to entering the study and have not recovered to baseline (except alopecia) or ≤ Grade 1 AEs, or deemed irreversible from the effects of prior cancer therapy. AEs > Grade 1 that are not considered a safety risk by the Sponsor and investigator may be allowed upon agreement with both, including residual neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of ADI-PEG 20 in combination with nab-Paclitaxel and Gemcitabine in Advanced Pancreatic Cancer | course of study - 1 year expected

CONTACTS AND LOCATIONS:
Overall Officials: Maeve Lowery, MD, Principal Investigator — Memorial Sloan-Kettering Cancer Center (MSKCC)
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States